CLINICAL TRIAL: NCT06351280
Title: Evaluation of Performance-based Functional Outcome Measures After Open Abdominal Surgery: a Comparison of Clinimetric Properties of Four Tools
Brief Title: Evaluation of Performance-based Functional Outcome Measures After Open Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Sana Nasir Zaidi
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Laparotomy
Keywords: Post operative laparotomy, cardiopulmonary functionality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functionality Assessment (Other): Each participant will be provided with an informed consent form detailing the purpose of the study. After obtaining written consent, baseline data will be collected, including demographic information, medical history, and any pre-existing conditions. The participants will then undergo the post-laparotomy interventions as described. Throughout the intervention period, data will be collected using the tools mentioned: 6 minute Walk Test, 5 Times Sit to Stand test, 2 Minute walk Test, and Timed Up and GO to determine any changes in their functionality and overall well-being on post operative day 1 and before discharge. For reliability, tests will be conducted twice a day with a minimum gap of 2 hours, both on day 1 and on the day of discharge.
  Interventions: Other: Standardised Physiotherapy Plan

INTERVENTIONS:
Other: Standardised Physiotherapy Plan — Single session of coached deep breathing and coughing exercises. 10 supervised slow flow deep breaths to total lung capacity with a 3-5 second end inspiratory hold completed with 2 end inspiratory sniffs. 2-3 supported coughs or huffs. Repeated for another set. Patients instructed to perform independently hourly. Assisted ambulation according to the following protocol:
  * Stage 1 of 2 minutes.
  * Stage 2 of 0-1 minute.
  * Stage 3 of 1 - 3 minutes.
  * Stage 4 of 3 - 6 minutes.
  * Stage 5 of 6 - 10 minutes.
  * Stage 6 of 10 - 15 minutes.
  * Stage 7 > 15 minutes. Total session time is the accumulative work time.

SUMMARY:
A laparotomy is a surgical technique, the increasing rate of this surgical interventions and the subsequent need to evaluate the post-surgical recovery and rehabilitation process comprehensively. This study aims to provide essential insights into the reliability, validity, and responsiveness of such tests, enabling healthcare professionals to make informed decisions about patient recovery progress and the optimization of rehabilitation protocols.

DETAILED DESCRIPTION:
The significance of this research lies in its potential to enhance the quality of care and patient outcomes, reduce healthcare costs, and contribute to evidence-based decision-making in postsurgical rehabilitation, ultimately improving the overall well-being of surgical patients. This study is to evaluate the clinimetric properties of four distinct tools designed for assessing performance-based functional outcomes following open abdominal surgery. 6 Minute Walk Test (6MWT), 5 Times Sit to Stand test (5T STS), 2 minute Walk test (2MWT), and Timed Up and GO (TUG)will be assessed to determine any changes in their functionality and overall well-being on day 2 and on day of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Post-laparotomy patients
* Hemodynamically stable
* Age between 30 to 60 years
* Ambulatory patients
* Patients score 1

Exclusion Criteria:

* Incidence of adverse events through hemodynamic and medication data.
* Diagnosed cognitive dysfunction.
* Diagnosed neurologic or musculoskeletal disease (excluding osteoarthritis) adversely affecting gait or weight-bearing.
* History of Orthostatic intolerance.
* History of recent fractures, blunt trauma emergency laparotomy, carcinoma.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
6MWT (Six-Minute Walk Test) | 1 week
  A submaximal exercise test called the 6MWT is used to measure aerobic capacity and endurance. This test's main goal is for the patient to walk as far as they can in six minutes.
  6MWT (Six-Minute Walk Test) A submaximal exercise test called the 6MWT is used to measure aerobic capacity and endurance. The distance (measured in meters) traveled during the six minutes allotted for the test determines the score.
5 Times Sit to Stand | 1 week
  The test can be used to track the course of an illness or the effectiveness of a therapeutic intervention in addition to providing useful information about a person's functional ability. The distance (measured in meters) traveled during the six minutes allotted for the test determines the score. Greater aerobic endurance and functional capacity are indicated by a longer distance
2MWT (Two-Minute Walk Test) | 1 week
  The 2MWT is a functional exercise test designed to evaluate an individual's aerobic capacity and endurance over a shorter duration compared to the 6MWT.
Timed Up and GO (TUG) | 1 week
  . It is designed to assess an individual's mobility and requires the participant to stand up from a seated position, walk a distance of three meters, turn around, walk back to the chair, and sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boden I, Sullivan K, Hackett C, Winzer B, Hwang R, Story D, Denehy L. Intensive physical therapy after emergency laparotomy: Pilot phase of the Incidence of Complications following Emergency Abdominal surgery Get Exercising randomized controlled trial. J Trauma Acute Care Surg. 2022 Jun 1;92(6):1020-1030. doi: 10.1097/TA.0000000000003542. Epub 2022 Jan 18. PMID 35609291
- [Background] . Li AM, Yin J, Yu C, Tsang T, So H, Wong E, et al. The six-minute walk test in healthy children: reliability and validity. 2005;25(6):1057-60. 16. Goldberg A, Chavis M, Watkins J, Wilson TJAc, research e. The five-times-sit-to-stand test: validity, reliability and detectable change in older females. 2012;24:339-44. 17. Cristina da Silva L, Danielli Coelho de Moraes Faria C, da Cruz Peniche P, Ayessa Ferreira de Brito S, Tavares Aguiar LJTiSR. Validity of the two-minute walk test to assess exercise capacity and estimate cardiorespiratory fitness in individuals after stroke: a cross-sectional study. 2023:1-10. 18. Bohannon RW, Wang Y-C, Gershon RCJAopm, rehabilitation. Two-minute walk test performance by adults 18 to 85 years: normative values, reliability, and responsiveness. 2015;96(3):472-7.